CLINICAL TRIAL: NCT04597710
Title: Precision Medicine for Liver Tumours With Quantitative Magnetic Resonance Imaging and Whole Genome Sequencing
Acronym: Precision1
Status: Active, not recruiting | Type: Observational
Sponsor: Perspectum (Industry)
Responsible Party: Sponsor
Other Study IDs: 20/PR/0222
Record Dates: First submitted 2020-10-13; First posted 2020-10-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Liver Cancer; Liver Metastasis Colon Cancer
Keywords: MRI; Surgery; Whole genome sequencing
MeSH Terms: conditions — Liver Neoplasms | interventions — Whole Genome Sequencing; Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Retention of histopathlogy samples: tumour and normal tissue; also serum, plasma and buffy coat, extracted DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: utility of whole genome sequencing (WGS) to aid clinical decision making in patients referred for liver resection — All participants will attend their planned outpatient surgery appointment.The consultant will document the intended treatment plan for each participant in line with their usual care pathway.Following this, participants will be required to attend three dedicated study visits:The results of the MRI scans from Study Visit 1 will be analysed into a LiverMultiScan report.A report will be sent to the consultant who will review their original documented care plan alongside the LiverMultiScan report.The consultant may update the intended care plan as a result of the LiverMultiScan report, in line with the device CE-marking.Any changes to the care plan will be documented.The patient will then undergo their planned treatment.The tumour explant will be collected and samples will be stored, transported and processed for genetic sequencing and digital histopathology.Study Visit 2 will be performed remotely 12 months following their planned treatment,where patient reported outcomes will be collected

SUMMARY:
This will be a prospective, observational, cohort study to determine the impact of integrated diagnostics using quantitative magnetic resonance imaging, whole genome sequencing and digital pathology on intended patient management for liver cancer patients referred for liver resection.

Participants with primary or secondary liver cancer will be recruited from Hampshire Hospitals NHS Foundation Trust in Basingstoke or Oxford University Hospitals NHSFoundation Trust in Oxford. The incidence of treatable liver tumours is on the rise globally, driven by obesity, viral hepatitis and metastases from colorectal cancers. Survival rates can be improved with optimised allocation of treatment options including surgical resection, radiofrequency ablation, embolisation, chemotherapy and targeted molecular therapies (including immunotherapy).

The key motivation of this study is to help patients access the most suitable treatment combinations, based on integrating clinical, radiological and genomic data. A similar integrated approach, integrating radiology and pathology, has been shown to improve outcomes in breast cancer care. Detailed pathologic analysis of the surgical specimen from breast carcinoma biopsy provides valuable feedback to the radiologist, establishes the completeness of surgical intervention, and generates predictive information for therapeutic decisions. Whole genome sequencing (WGS) has discovered cancer driver mutations and the complex molecular profile of liver cancer. In many metastatic solid tumours, WGS has been used to identify a significant patient population (31%) who present with a biomarker that predicts sensitivity to a drug and lacked any known resistance biomarkers for the same drug. Identifying which patients possess druggable mutations will allow clinicians to make the optimal treatment decisions. The next challenge is integrating WGS into scalable clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age and older willing and able to give informed consent to participate in the study
* Patients being considered for liver resection for primary or secondary liver cancer.

Exclusion Criteria:

* The participant may not enter the study with any known contraindication to magnetic resonance imaging (including but not limited to pregnancy, a pacemaker or other metallic unfixed implanted device, metallic fragments, extensive tattoos, severe claustrophobia).
* Any other cause, including a significant underlying disease or disorder which, in the opinion of the investigator, may put the participant at risk by participating in the study or limit the participant's ability to participate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The primary endpoint of the study is an evaluation of the number of patients for whom clinically actionable data is provided by whole genome sequencing.
  Based on the following information, we will aim to recruit 200 patients from HHFT and expect to observe at least a 25% change in intended clinical management (at 95% confidence interval).
  * A recent study using whole-genome analyses of metastatic solid tumours identified 31% of patients who present with a biomarker that predicts sensitivity to a drug and lacked any known resistance biomarkers for the same drug.
  * The primary end-point can be achieved with only the first study visit, and so no drop-out is expected.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients for whom clinically-actionable data is provided by whole genome sequencing at the time of surgery. | 36 months
  This will be evaluated retrospectively, with clinically-actionable data defined as data which would result in a clinician choosing a different medical intervention to the current standard of care.

SECONDARY OUTCOMES:
Proportion of patients for whom clinically-actionable data is provided by LiverMultiScan. | 36 months
  . To determine the utility of quantitative multiparametric MRI with LiverMultiScan to aid clinical decision making in patients referred for liver resection.
Correlation of computationally-derived digital pathology results with human pathologist assessments of the tumour and non-tumour tissue, along with assessment of intra- and inter-rater variability. | 36 months
  To compare computationally-derived digital pathology results with human pathologist assessments of the tumour and non-tumour tissue.
Correlation of MR measurements of steatosis and fibroinflammation with digital pathology and human pathology. | 36 months
  To compare histopathological assessments of liver fat and fibroinflammation with quantitative MRI metrics (cT1, PDFF)
Performance of WGS and LiverMultiScan for predicting post-surgery length of stay in hospital, post-operative liver function, 1-year mortality and recurrence rates. | 36 months
  To evaluate the long term outcomes and recurrence rates and recurrence patterns of patients as it relates to imaging and whole genome sequencing.
Proportion of patients for whom actionable biomarkers of drug sensitivity are identified with WGS. | 36 months
  To evaluate whether whole genome sequencing enables better stratification of patients prior to surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Rajarshi Banerjee, Principal Investigator — Perspectum Ltd
Locations (1):
- Basingstoke and North Hampshire Hospital, Basingstoke, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Welsh FK, Connell JJ, Kelly M, Gooding S, Banerjee R, Rees M. Precision medicine for liver tumours with quantitative MRI and whole genome sequencing (Precision1 trial): study protocol for observational cohort study. BMJ Open. 2022 Apr 5;12(4):e057163. doi: 10.1136/bmjopen-2021-057163. PMID 35383076